CLINICAL TRIAL: NCT01976676
Title: Comparison of the Effect of Folic Acid and 5-methyltetrahydrofolate (5MTHF) on Serum Folate and Homocysteine Levels, and Abortion Rates in Women Suffering From Recurrent Abortion
Brief Title: Folic Acid vs 5-methyltetrahydrofolate (5MTHF) in Recurrent Abortion
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Associate Prof, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1157
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Recurrent Abortion
MeSH Terms: conditions — Abortion, Habitual | interventions — 5-methyltetrahydrofolate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-methyltetrahydrofolate (Experimental): 1 mg 5-methyltetrahydrofolate per day
  Interventions: Dietary Supplement: 5-methyltetrahydrofolate
- folic acid (Active Comparator): 1 mg Folic acid per day
  Interventions: Dietary Supplement: folic Acid

INTERVENTIONS:
Dietary Supplement: 5-methyltetrahydrofolate
  Arms: 5-methyltetrahydrofolate
Dietary Supplement: folic Acid
  Arms: folic acid

SUMMARY:
Recent data indicates that 5 methyltetrahydrofolate (5MTHF) can reduce serum homocystein level more efficiently than folic acid. On the other hand, folic acid is currently an important part of treatment in idiopathic recurrent abortion. There is no study comparing the effectiveness of these supplements in the treatment of recurrent abortion. The aim of this study is to compare the efficiency of these two agents in the treatment of recurrent abortion. In this study, patients with idiopathic recurrent abortion, referring to Avicenna clinic will be randomly allocated into two groups of those taking either folic acid (5 mg) or 5 MTHF (5mg) from 8 weeks prior to conception until the 20th week of pregnancy. The serum level of folate, homocystein, and ongoing pregnancy will be analysed and compared in the two groups.

ELIGIBILITY:
Inclusion criteria:

* Willing to participate in the study and filling out the informed consent form,
* History of 3 or more idiopathic abortion,
* the last abortion should be more than 6 months ago,
* no history of consumption of folate supplements or high folate containing foods during last 6 months,
* All previous abortions should be idiopathic without any anatomic, cytologic, hormonal, septic pathologic finding,
* no special diets

Exclusion Criteria:

* elective or induced abortion, molar or ectopic pregnancies,
* presence of any malignancy, chromosomal abnormality, uterine abnormality, Thyroid, kidney, or liver dysfunction, Glucose intolerance, seizure,
* Alcohol or drug abuse,
* Taking any drug affecting homocystein metabolism,
* not following the study protocol.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy on the 20th week of gestational age | 20th week of gestational age

SECONDARY OUTCOMES:
serum concentration of folate | at the weeks 0 and 8 of the study, and weeks of 4, 8, 12, and 20th gestational age
Serum concentration of Homocystein | at the weeks 0 and 8 of the study, and weeks of 4, 8, 12, and 20th gestational age

REFERENCES:
- [Derived] Hekmatdoost A, Vahid F, Yari Z, Sadeghi M, Eini-Zinab H, Lakpour N, Arefi S. Methyltetrahydrofolate vs Folic Acid Supplementation in Idiopathic Recurrent Miscarriage with Respect to Methylenetetrahydrofolate Reductase C677T and A1298C Polymorphisms: A Randomized Controlled Trial. PLoS One. 2015 Dec 2;10(12):e0143569. doi: 10.1371/journal.pone.0143569. eCollection 2015. PMID 26630680